CLINICAL TRIAL: NCT00957788
Title: Safety and Feasibility Study of NST - 001 in Inner Ear Using Neuroject Injection Set for the Treatment of Tinnitus
Brief Title: Safety Study for NST-001 and the Neuroject Injection Set to Treat Tinnitus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroSystec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NST-CP-02
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2011-06

CONDITIONS: Tinnitus
Keywords: tinnitus; acouphenes; ear; ringing; buzzing; roaring; hissing; clicking
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 0 (Experimental)
  Interventions: Drug: NST-001
- Cohort 1 (Experimental)
  Interventions: Drug: NST-001
- Cohort 2 (Experimental)
  Interventions: Drug: NST-001
- Cohort 3 (Experimental)
  Interventions: Drug: NST-001

INTERVENTIONS:
Drug: NST-001 — Comparison of different dosages of drug.

SUMMARY:
This research study involves an experimental drug (NST_001) and a delivery system. The main purpose of this research study is to investigate the safety of NST-001, delivered directly to the inner ear for the treatment of tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to provide voluntary consent.
* Severe tinnitus in one ear that began no more than ten years ago.
* Ear to be treated must be deaf or have profound hearing loss.
* Subjects with cardiac disease or hypertension, must have stable disease for at least 6 months.
* Subject must have intact cochlear nerve on the ear to be treated.
* Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods as recommended by the study physician.

Exclusion Criteria:

* Current diagnosis of bilateral tinnitus.
* Current diagnosis or history of pancreatitis.
* Females that are pregnant or lactating.
* Use of investigational drugs within the previous 30 days.
* History of drug dependency or other substance abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Subjects will be followed for identification and frequency of drug or procedure-related adverse events. | At each follow-up visit.

SECONDARY OUTCOMES:
Observe any effect on tinnitus as determined by the visual analog scale, subject tinnitus diary, and investigator interview. | At each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Frachet, MD, Principal Investigator — Hôpital Avicenne; Pierre Garin, MD, Study Director — Cliniques Universitaries U.C.L.
Locations (2):
- Cliniques Universitaries U.C.L., Mont-Godinne, Belgium
- Hôpital Avicenne, Bobigny, Cedex, France